CLINICAL TRIAL: NCT07190651
Title: Development of a New Remote Monitoring Model for Patients With HR+HER2- Breast Cancer in Treatment With CDK4/6 Inhibitors and Hormone Therapy
Acronym: VIRTUOSA
Status: Not yet recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Paris Ida, Head of Unit, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: ID 7960
Record Dates: First submitted 2025-09-17; First posted 2025-09-24 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer; CDK4/6 Inhibitor
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women with advanced HR-positive/Her2-negative Breast Cancer: Women with advanced HR-positive/Her2-negative Breast Cancer (BC) who have completed at least 2 cycles of a first-line therapy with CDK4/6i + hormone therapy and are currently on treatment.
  Interventions: Other: Home questionnaire

INTERVENTIONS:
Other: Home questionnaire — Administration of a questionnaire at each 28-days cycle, to select patients who need to access to hospital for clinical visit during treatment with CDK4/6i + hormone therapy for advanced breast cancer.

SUMMARY:
This study aims to develop and prospectively validate a questionnaire to select patients with breast cancer who need to access to hospital for clinical visit during treatment with CDK4/6i, to improve patients' quality of life and reduce burden of hospital accesses.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent.
* Age ≥18 years old
* Histologically or cytologically documented diagnosis of HR+, HER2-negative breast cancer based on local laboratory results and who are not amenable to resection or radiation therapy with curative intent. HR+ tumor is defined as ER and/or PgR expression in greater than 1% of tumor cells. HER2-negative breast cancer is defined as a negative in situ hybridization test or an immunohistochemistry (IHC) status of 0 or 1+. If IHC is 2+, a negative in situ hybridization (FISH, CISH, or SISH) test is required to confirm the HER2-negative status (based on the most recently analyzed tissue sample tested by a local laboratory).
* Currently on treatment and have received ≥ 2 months of CDK4/6i + hormone therapy as their initial endocrine based treatment for their metastatic disease in concordance with local CDK4/6i label or treatment guideline.
* No evidence of clinical or radiological disease progression per investigator assessment.
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) ≤2.

Exclusion Criteria:

* History of significant neurological or psychiatric disorders that would prohibit the understanding and giving of informed consent.
* Patient has a concurrent invasive malignancy and /or is concurrently using other anti-neoplastic therapy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with advanced HR-positive/Her2-negative Breast Cancer (BC) who have completed at least 2 cycles of a first-line therapy with CDK4/6i + hormone therapy and are currently on treatment.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Concordance between the results of the questionnaire and the clinical examination of the patients. | 12 months
  This study will validate a questionnaire to select patients who need to access to hospital for clinical visit during treatment with CDK4/6i + hormone therapy for advanced breast cancer. Concordance between the results of the questionnaire (3 flags) and the clinical examination of the patients will be evaluated.

IPD SHARING:
Plan to Share IPD: No